CLINICAL TRIAL: NCT03087604
Title: Loss of Resistance With Nerve Stimulation Versus Loss of Resistance Alone; Effect on Success of Thoracic Epidural Placement.
Brief Title: Loss of Resistance, w/wo Stimulation, For Epidural Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00039522
Record Dates: First submitted 2017-03-03; First posted 2017-03-22 (Actual); Results first posted 2018-11-23 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia
Keywords: epidural catheter placement
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Solutions; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: As the patient will be sedated during epidural catheter placement, they will be blinded to their treatment arm. The investigator that determines if the epidural was successful placed will also be blinded to the patient's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional Technique Group (Active Comparator): In the traditional loss of resistance technique group, the epidural catheter will be placed after achieving loss of resistance to air. After placement of the catheter a standard test dose of 3+2 ml of 1.5% lidocaine with 1:200,000 epinephrine will be administered.Solution for Thoracic epidural block.
  Interventions: Procedure: Thoracic epidural block; Drug: Solution For Thoracic epidural block
- Electric Stimulation Group (Experimental): In the electrical stimulation group, following the location of the epidural space with a loss of resistance technique (using air), nerve stimulation will be utilized to elicit a myotomal contraction of the abdominal or thoracic wall. After placement of the catheter a standard test dose of 3+2 ml of 1.5% lidocaine with 1:200,000 epinephrine will be administered.Solution for Thoracic epidural block.Thoracic epidural block with Electrical Nerve stimulation
  Interventions: Procedure: Thoracic epidural block; Procedure: Electrical Nerve stimulation; Drug: Solution For Thoracic epidural block

INTERVENTIONS:
Procedure: Thoracic epidural block — Thoracic epidural block with epidural placed with a loss of resistance technique alone.
Procedure: Electrical Nerve stimulation — In the electrical stimulation group, following the location of the epidural space with a loss of resistance technique (using air), nerve stimulation will be utilized to elicit a myotomal contraction of the abdominal or thoracic wall.stimulating peripheral nerve catheters(19 Ga. x 90 cm StimuCath® Continuous Nerve Block Catheter with SnapLock™ Adapter (Arrow by Teleflex Medical, Morrisville, NC), and stimulation will be achieved using a B Braun Stimuplex HNS12 Nerve Stimulator product id 4892098.
  Arms: Electric Stimulation Group
Drug: Solution For Thoracic epidural block — Dose of 3+2 ml of 1.5% lidocaine with 1:200,000 epinephrine
  Other Names: Lidocaine; Epinephrine

SUMMARY:
The purpose of this randomized, observer-blinded, investigative trial is to determine if the use of electrical stimulation, compared to the traditional loss of resistance technique alone, improves the success rate of epidural catheter placement at an academic teaching institution.

DETAILED DESCRIPTION:
All subjects will receive a thoracic epidural catheter placement at the level appropriate for their surgery and will be randomized to either have the epidural placed with a loss of resistance technique alone or loss of resistance technique with confirmation by nerve stimulation. In the traditional loss of resistance technique group, the epidural catheter will be placed after achieving loss of resistance to air. In the electrical stimulation group, following the location of the epidural space with a loss of resistance technique (using air), nerve stimulation will be utilized to elicit a myotomal contraction of the abdominal or thoracic wall. Nerve stimulation will be started at a pulse width of 0.3 ms and a frequency of 1 Hz and a current of 0.2mA.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing intra-thoracic or intra-abdominal procedures that normally would receive thoracic epidurals for post-operative analgesia will be eligible.

Exclusion Criteria:

* Subjects with contraindications to regional anesthesia:
* history of allergy to amide local anesthetics
* presence of a progressive neurological deficit
* patients that are on anticoagulant medications that prohibit placement of an epidural
* Systemic infection
* Infection at the site of placement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Dobson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- WakeForestUBMC, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dobson SW, Weller RS, Edwards C, Turner JD, Jaffe JD, Reynolds JW, Henshaw DS. A randomized comparison of loss of resistance versus loss of resistance plus electrical stimulation: effect on success of thoracic epidural placement. BMC Anesthesiol. 2022 Feb 9;22(1):43. doi: 10.1186/s12871-022-01584-x. PMID 35139802

RESULTS

PARTICIPANT FLOW:
Groups:
- Electric Stimulation Group: In the electrical stimulation group, following the location of the epidural space with a loss of resistance technique (using air), nerve stimulation will be utilized to elicit a myotomal contraction of the abdominal or thoracic wall. After placement of the catheter a standard test dose of 3+2 ml of 1.5% lidocaine with 1:200,000 epinephrine will be administered.Solution for Thoracic epidural block.Thoracic epidural block with Electrical Nerve stimulation
  Thoracic epidural block: Thoracic epidural block with epidural placed with a loss of resistance technique alone.
  Electrical Nerve stimulation: In the electrical stimulation group, following the location of the epidural space with a loss of resistance technique (using air), nerve stimulation will be utilized to elicit a myotomal contraction of the abdominal or thoracic wall.stimulating peripheral nerve catheters
Period: Overall Study
Arm/Group | Traditional Technique Group | Electric Stimulation Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Technique Group | Electric Stimulation Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12.6) | 60.4 (15.4) | 61.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 31 | 23 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 45 | 46 | 91
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Placement of a Thoracic Epidural
Description: will be determined by the detection of a loss of sensation to cold (ice) in at least two contiguous dermatomal levels, 15 minutes after administration of a test dose of lidocaine through the epidural catheter. If a loss of cold sensation is found, then the epidural placement will be classified as successful. If no loss of cold sensation is found, then the epidural placement will be classified as unsuccessful.
Time Frame: 15 minutes after administration of a test dose of lidocaine
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Technique Group | Electric Stimulation Group
Number analyzed (Participants) | 50 | 50
Participants | 41 | 45

2. Secondary Outcome: Time Required to Place the Epidural Catheter
Description: The time required to place the epidural catheter will be recorded
Time Frame: From the initiation of procedure to end of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Traditional Technique Group | Electric Stimulation Group
Number analyzed (Participants) | 50 | 50
minutes | 33.9 (12.8) | 24.0 (8.0)

3. Secondary Outcome: Number of Thoracic Spine Levels Attempted
Description: the number of thoracic spine levels attempted will be recorded
Time Frame: Thirty minutes after start of procedure.
Population: No data collected
Arm/Group | Traditional Technique Group | Electric Stimulation Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 30 minutes
Arm/Group | Traditional Technique Group | Electric Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT03087604/Prot_SAP_000.pdf